CLINICAL TRIAL: NCT01379677
Title: Diagnosis of Coronary Artery Disease With Rubidium-82 PET and Technetium-99m-MIBI SPET: A Head to Head Comparison, Versus Coronary CT Angiography
Brief Title: Rubidium-82 PET and Tc-99m-MIBI SPET: A Head to Head Comparison
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009Rb82UK; 2009-016645-25 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-23 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Myocardial perfusion imaging; Rubidium; Technetium
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rubidium-82; Sodium Pertechnetate Tc 99m

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): This is an Head to Head Comparison between Rubidium-82 PET and Tc-99m-MIBI SPET with CTA as gold standard. All the patients will undergo the three imaging protocols.
  Interventions: Drug: Rubidium-82; Drug: Sestamibi. reconstitution with sodium pertechnetate (99mTc)

INTERVENTIONS:
Drug: Rubidium-82 — Maximum dose allowed per injection: 2200 MBq Maximum cumulated dose allowed per examination: 4400 MBq Intravenous Use
  Other Names: CardioGen-82
Drug: Sestamibi. reconstitution with sodium pertechnetate (99mTc) — Maximum dose allowed per injection: 1000 MBq Intravenous Use
  Other Names: Technescan MIBI

SUMMARY:
The main purpose of this study is to compare myocardial perfusion imaging using Rubidium-82 PET with Tc-99m-MIBI SPET, in the evaluation of significant Coronary Artery Disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* Referred for scintigraphy to assess myocardial ischaemia
* Ability to give informed written consent.

Exclusion Criteria:

* Impaired capacity to consent
* Pregnancy, or breastfeeding
* Allergy to iv contrast
* Renal failure
* Severe Uncontrolled asthma
* Claustrophobia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The specificity of detecting significant coronary artery disease (as defined as being >70% stenosis, on coronary CT angiography) | Up to 2 days
  The primary objective is to compare PET vs. SPET, with the primary outcome being the specificity of detecting significant coronary artery disease (as defined as being >70% stenosis, on coronary CT angiography).

SECONDARY OUTCOMES:
Evaluate any difference in the clinical interpretation of the Rubidium-82 PET and Tc-99m-MIBI SPET images. | Up to 2 days
Evaluate any difference in "Percentage myocardium" that is hypoperfused, between Rubidium-82 PET and Tc-99m-MIBI SPET. | Up to 2 days
Evaluate any difference in image quality, artefacts and interpretative confidence between Rubidium-82 PET and Tc-99m-MIBI SPET. | Up to 2 days
Evaluate any adverse events or reactions, during Rubidum-82 or Tc-MIBI administration. | Up to 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Leon Menezes, Dr., Principal Investigator — University College Hospital London NHS Foundation Trust
Locations (1):
- University College Hospital London NHS Foundation Trust, London, London, United Kingdom